CLINICAL TRIAL: NCT07300631
Title: OASIS: SpaceOAR PoSt - Market Registry Study: Assessing the Safety & Acceptability of SpaceOAR Use With Prostate Radiotherapy
Brief Title: SpaceOAR Post-Market Registry Study
Acronym: OASIS
Status: Recruiting | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Clinique Pasteur Toulouse (Other); Sheffield Hallam University (Other)
Responsible Party: Sponsor
Other Study IDs: STH22555; IRAS Project ID: 341038 (Other: HRA)
Record Dates: First submitted 2025-11-19; First posted 2025-12-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer Patients Treated by Radiotherapy
Keywords: rectal spacer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- All participants: Participants receiving prostate cancer care in the UK and France
  Interventions: Device: SpaceOAR / SpaceOAR Vue hydrogel system

INTERVENTIONS:
Device: SpaceOAR / SpaceOAR Vue hydrogel system — Space OAR/SpaceOAR Vue Systems are biodegradable medical devices that are implanted between the prostate and rectum to temporarily move part of the rectal wall away from the prostate during radiation therapy for prostate cancer.

SUMMARY:
Recently, concerns have been raised by regulators that there is little data about the long-term safety of rectal hydrogel spacers for use in conjunction with radiotherapy treatment for prostate cancer. To address this, this study will collect data about the short-term side-effects and long-term safety of SpaceOAR and SpaceOAR Vue rectal hydrogel spacers in men who receive them in the UK and France. Men who have agreed to receive these spacers as part of their standard medical care will be asked to take part in the study whereby data about their treatment and health will be collected from their medical records and from members of the clinical team who deliver their treatment. Additionally, men will be asked to consent to completing questionnaires about their experiences of side effects from their treatment. Further information will be collected about their clinical characteristics before they receive a spacer, the physician-rated clinical performance of the spacer insertion procedure, their radiotherapy treatment plan and details of the other treatments they are also receiving which could influence the types and extent of side effects they experience. Data collection will span eight time points: pre-spacer insertion, spacer insertion, the start of radiotherapy, post-radiotherapy follow-up, 6-month follow-up, 12-month follow-up, 24-month follow-up & 36-month follow-ups. Outside of these timepoints treatment-related adverse event data will be concurrently reported and collated. Participants' treatments will not be changed as a result of their participation in this study. Data from this study will be used to summarise the characteristics of this study population, physicians' perceptions of the spacer implantation procedure, the radiotherapy treatments plans made, and the types, extent and timing of treatment-related adverse events and side effects.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a clinical diagnosis of prostate cancer planned to undergo treatment with curative intent at selected sites in the UK & France subject to a SpaceOAR being used as usual care.
* Aged 18 years old or above.
* Patients who agrees to participate and has been deemed by their medical team to have capacity to provide;

  * verbal, informed consent over telephone as documented on the study informed consent form by the Researchers (UK only)
  * written, informed consent by signature of the study informed consent form (France only)
* Patient covered by social security scheme (France only)

Exclusion Criteria:

- Patients lacking the capacity to provide;

* informed consent as documented on the study informed consent form by the - Researchers (UK only)
* written, informed consent by signature of the study informed consent form (France only)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with prostate cancer having radiotherapy with curative intent and having a SpaceOAR as part of standard care.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Short-term safety of SpaceOAR/SpaceOAR Vue systems. | 30 days post-implantation
  Proportion of subjects experiencing any of the following within 30 days post-implantation of SpaceOAR/SpaceOAR Vue hydrogel, as adjudicated by the Independent Clinical Events Committee:
  * Symptoms (PROMs): Measured using validated patient-reported outcome questionnaires. A subject is counted if any PROM score exceeds the predefined threshold for clinically significant symptoms.
  * Adverse Events (CTCAE v5.0): Measured as the occurrence of any adverse event graded per CTCAE v5.0.
  * Abnormal Imaging (MRI/CT): A subject is counted if any abnormality is confirmed by radiology review.
    * The study instruments in the French population with include Grade 1 and above events (CTCAEv5.0)
  * Unit of Measure: Percentage of subjects (%)
  * Each category will be reported separately.
Long-Term Safety of SpaceOAR/SpaceOAR Vue Systems | Up to 3 years post-radiation therapy
  Proportion of subjects experiencing Grade ≥2 gastrointestinal or anorectal toxicity (per CTCAE v5.0) within 3 years after completion of radiation therapy.
  * The study instruments in the French population with include Grade 1 and above events (CTCAEv5.0)
  • Unit of Measure: Percentage of subjects (%)

SECONDARY OUTCOMES:
Proportion of subjects with Grade 2* & above; gastrointestinal, anorectal, genitourinary toxicity at 12, 24 & 36 months. | 12, 24, and 36 months post-radiation therapy
  Proportion of subjects experiencing Grade ≥2 toxicity (as per CTCAE v5.0) in gastrointestinal, anorectal, or genitourinary systems at 12, 24, and 36 months post-radiation therapy.
  • Unit of Measure: Percentage of subjects (%) Note: For French population, Grade ≥1 events will also be included.
Physician rating of SpaceOAR/SpaceOAR Vue of Placement Difficulty | At time of implantation
  Rated on a Likert scale (1 = very difficult, 5 = very easy) immediately after procedure.
  Unit of Measure: Mean Likert score
Patient Perception of SpaceOAR/SpaceOAR Vue Procedure Compared to Prostate Biopsy | Within 30 days post-procedure
  Measured using a structured questionnaire comparing perceived discomfort and acceptability relative to prostate biopsy.
  • Unit of Measure: Percentage of subjects reporting "less discomfort," "similar," or "more discomfort
Overall Mortality and Cause of Death | Up to 36 months
  Number and proportion of subjects who die during the study period, with cause adjudicated by Independent Clinical Events Committee.
  • Unit of Measure: Number of deaths and percentage (%)
Selection Criteria for SpaceOAR/SpaceOAR Vue Placement | At enrolment
  Analysis of baseline clinical and demographic factors associated with successful placement.
  • Unit of Measure: Descriptive statistics (frequency, percentage)
Time to Onset of Grade ≥2 Gastrointestinal, Anorectal, and Genitourinary Toxicity | Up to 36 months
  Measured as time (in months) from radiation therapy completion to first occurrence of Grade ≥2 toxicity (per CTCAE v5.0).
  • Unit of Measure: Median time to onset (months)
Impact of treatment on bowel function, urinary function, sexual function and overall quality of life as measured by EPIC-26 | Baseline, 12, 24 and 36 months
  The EPIC-26 questionnaire is a preeminent tool extensively characterised to measure health-related quality of life in men with localised prostate cancer across specific domains
  * Urinary function
  * Bowel function
  * Sexual function
  * Effects of hormone treatment Scores range from 0-100, with higher scores indicating better function or quality of life.
  Unit of Measure: Mean score change from baseline (points)
Impact of treatment on bowel function, urinary function, sexual function and overall quality of life as measured by IPSS | Baseline, 12, 24 and 36 months
  International Prostate Symptom Score (IPSS). IPSS assesses urinary voiding symptoms and bother.
  For voiding symptoms, a score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms, and the urinary bother scale ranges from 0 (Delighted) to 6 (Terrible).
  Unit of Measure: Mean score change from baseline (points)
Impact of treatment on bowel function as measured by Vaizey incontinence score | Baseline, 12, 24 and 36 months
  The Vaizey Incontinence Score is a general-purpose scale for faecal incontinence that ranges from 0 to 24 with higher scores representing worst incontinence.
  Unit of Measure: Mean score change from baseline (points)
Impact of concomitant prostate cancer treatment usually Androgen Deprivation Therapy (ADT) on the lives of participants as measured by The Symptom Index | Baseline, 12, 24, 36 months
  The Symptom Index is an un-validated questionnaire which has been developed to capture the impact of the side effects of concomitant prostate cancer treatment (usually ADT} on the lives of participants. The questions capture the quality of life using the scale: 0 - 4, with higher scores indicating worse symptoms or quality of life.
  Unit of measure: Mean score change from baseline (points)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Rosario, Study Chair — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (8):
- France (3):
  - CHU de Brest, Brest
  - Clinique Pasteur, Toulouse
  - Centre de cancérologie Les Dentellières, Valenciennes
- United Kingdom (5):
  - Chesterfield Royal Hospital, Chesterfield
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Royal Free Hospital, London
  - Maidstone & Tunbridge Wells NHS Trust, Maidstone
  - Norfolk & Norwich University Hospital NHS Foundation Trust, Norwich

IPD SHARING:
Plan to Share IPD: No